CLINICAL TRIAL: NCT04188002
Title: A Web-based Tailored Health Behavior Intervention for Breast and Colon Cancer Survivors (eWellness)
Acronym: eWellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 16-1897
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Nutrition; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single institution, randomized clinical trial designed to evaluate a four week web-based tailored health behavior intervention in breast and colon cancer survivors.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Fruit and Vegetable (Other): Participants in this arm will receive usual care.
  Interventions: Other: Usual Care
- Physical Activity Intervention (Other): Participants in this arm will be encouraged via tailored newsletters and email/or text reminders to improve diet and physical activities.
  Interventions: Behavioral: Intervention Physical Activity

INTERVENTIONS:
Behavioral: Intervention Physical Activity — 4 tailored newsletters focused on improving healthy diet and physical activity delivered at weekly intervals.
  Arms: Physical Activity Intervention
Other: Usual Care — 4 non-tailored newsletters focused on issues relevant to cancer survivors (e.g. returning to work)
  Arms: Control - Fruit and Vegetable

SUMMARY:
The primary objective of this study is to compare the differences in fruits and vegetable intake and physical activity from pre- to post- study between the intervention and control groups (i.e. the difference in differences). The study involves the use of web-based educational materials over a four week period. The investigators hypothesize that those in the intervention group will show a greater increase in fruit and vegetable intake and engage in more physical activity than those randomized to the control group. Eligible breast and colorectal cancer survivors from the UNC Health Registry/Cancer Survivorship Cohort (UNC HR/CSC) will be selected, consented, and randomized to either the intervention or control group. Both groups will fill out baseline surveys. The intervention group will receive a total to 4 newsletters for 4 weeks and at the beginning of week 5, they will asked to complete the follow-up survey online. The intervention newsletters focus on increasing physical activity and healthy diets. The control group will receive 4 newsletters in the same time frame as the intervention. The focus of the control group's newsletters will be on topics relevant to cancer survivors (e.g. getting back to work after treatment, managing finances) but will not focus on physical activity or diet. All contact with participants will take place online (i.e. surveys and newsletter delivery) from the study web site.

DETAILED DESCRIPTION:
This study is adapted from the WATCH (Wellness for African Americans Through Churches) Project. WATCH was a randomized trial among 587 African American members of 12 rural North Carolina churches that demonstrated the effectiveness of a mailed tailored print and video intervention consisting of four individually tailored newsletters and targeted videos to improve diet and physical activity behaviors: there were significant improvements in fruit and vegetable consumption (0.6 servings) and recreational physical activity (2.5 MET-hours per week), and a non-significant decrease in fat intake in the intervention churches. The overall goal of this application is to conduct a study (called "eWellness") to investigate whether the WATCH tailored print messages and videos can be effectively and efficiently disseminated to a different population (breast and colon cancer survivors) and using a different delivery channel (electronic technology via the internet and world wide web.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* primary language is English
* histologically confirmed stage 1-111A invasive breast cancer or stage 1-3 colorectal cancer
* between at least 6 months to 5 years since completion of all primary cancer treatments (e.g. surgery, radiation, chemotherapy with the exception of women on adjuvant Herceptin therapy)
* have access to the internet; have an email and/or cell phone (to accept text message reminders from the study).

Exclusion criteria:

Include women that may be pregnant and anyone that is/has:

* A history of another cancer (exception for non-melanoma skin cancers)
* Self-reported comorbidities that would preclude engaging in physical activity safely (e.g. functional limitations or symptomatic cardiovascular or pulmonary disease)
* Plans or scheduled for major surgery (including breast reconstruction) during the intervention time frame
* Any psychiatric illness that would make it difficult to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Mean Fruit and Vegetable Score | Month 6
  Fruit and vegetable consumption will be adapted from a 35-item measure used in a trial for US Blacks adapted from a 35-item measure for US Southern blacks that measures frequency of intake during the previous month. Score measures can range from 2-24. Positive or better outcomes are reflected by higher mean fruit and vegetable scores.
Summary Fruit and Vegetable Score | Month 6
  The frequency of fruit and vegetable intake will be measured during the previous month, using a 2-item measure (How many servings of fruits do you eat each day?) and a similar question for vegetables that assesses usual vegetable intake. Scores can range from 0-N with higher scores indicating more fruit and/or vegetable intake.
Metabolic Equivalent Task Hours (METs) for Physical Activity | Month 6
  Moderate to physical activity will be assessed and frequency of different types of activity, with response options of: don't do, 1-3 times/month, 1-2 times/week, 3-4 times/week, or 5 or more times/week. Items include various types of activities gathered from an 11-item instrument modified for cultural appropriateness from a previous study. For each activity, participants estimate duration as either <20 minutes or 20 or more minutes per session. Physical activity is then calculated in terms of metabolic equivalent task hours (METs) per week. MET values for energy expenditure were assigned to each activity based on validated instruments.21 MET-hours are computed by multiplying frequency times duration (converted to hours/week) times the MET value. Reported physical activity time can range from 0 minutes - 6 hours or more for reported sedentary behaviors. Higher reported values equate to better reported outcomes of increased physical activity for participants.

SECONDARY OUTCOMES:
Recruitment rate | Month 6
  Recruitment rate is defined as the number of screened participants that meet eligibility criteria divided by the number of individuals screened.
Percentage of Participants Completing the Intervention and Follow-Up Assessments | Month 6
  Retention
Number of Newsletters Read/Downloaded | Month 6
  Participant Adherence
Program Process Evaluation | 6 months
  This will be assessed with process evaluation questions at follow-up survey and metrics of website use (e.g. number of times visiting site). Questions will ask about participants' perceptions and experiences with the intervention and may provide valuable information about how to modify the programs for future use in this population. Measures will be adapted from those used in our previous studies and assess ease of use, intervention instructions and length, attractiveness, perceived personal relevance, recall, credibility, novelty, and usefulness for making healthy changes, and satisfaction with intervention components. Higher values will represent better outcomes for program process evaluation.
Number of Times Visiting the Site | 6 months
  An evaluation of website metrics will be conducted to assess program acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Carmina Valle, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Resnicow K, Morabia A. The relation between body mass index and plasma total cholesterol in a multiracial sample of US schoolchildren. Am J Epidemiol. 1990 Dec;132(6):1083-90. doi: 10.1093/oxfordjournals.aje.a115751. PMID 2260540